CLINICAL TRIAL: NCT00001789
Title: An Open-Label, Multiple-Dose Study to Evaluate the Efficacy, Safety and Pharmacokinetics of BG9588 (Anti-CD40L Antibody) in Subjects With Proliferative Lupus Glomerulonephritis (SLE-GN)
Brief Title: BG9588 (Anti-CD40L Antibody) to Treat Lupus Nephritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990133; 99-AR-0133
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Glomerulonephritis, Membranoproliferative; Lupus Nephritis
Keywords: Autoantibody; Autoimmunity; Inflammation; Kidney; Lymphocyte; Proliferative Lupus Glomerulonephritis; SLE-GN
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative; Lupus Nephritis; Autoimmune Diseases; Inflammation

INTERVENTIONS:
Drug: BG9588

SUMMARY:
The purpose of this study is to investigate whether the experimental drug BG9588 can be used to treat lupus nephritis more effectively and with less toxicity than standard treatments, including cyclophosphamide (Cytoxan), azothioprine (Imuran) and prednisone.

The body's immune system naturally produces antibodies to fight foreign substances like bacteria and viruses. In autoimmune diseases like lupus, however, the body makes antibodies that attack its own tissues, causing inflammation and organ damage. Lupus antibodies attack and damage kidney cells. BG9588 can interfere with the production of these antibodies, and therefore, may lessen kidney damage in people with lupus nephritis.

This study will look at: how BG9588 enters and leaves the blood and body tissue over time; adverse effects of the drug; and whether treatment with BG9588 can result in less kidney damage than other therapies.

Study patients will be receive a 30-minute infusion of BG9588 into a vein every two weeks for three doses and then once every 28 days for four doses. Patients' steroid dosage may be tapered; individual adjustments will be made as required.

Patients screened for the study will undergo a physical examination, medical history, various blood and urine tests, as well as complete a quality of life questionnaire. Results of a previous kidney biopsy and chest X ray are also required. Many of these tests will be repeated throughout the study.

In a previous animal study, BG9588 treatment of mice with lupus nephritis improved their disease and survival.

DETAILED DESCRIPTION:
Studies in animals and humans with lupus nephritis have demonstrated that essential role of CD40 ligand/CD40 interaction in the production of pathogenic autoantibodies. Anti-CD40L antibody treatment of mice with lupus nephritis ameliorates disease and improves survival. BG9588 is a recombinant humanized monoclonal antibody that specifically binds to CD40 ligand (CD40L) expressed on the surface of activated T lymphocytes and thereby blocks the CD40L/CD40 interaction between T and B cells that is required for the initiation for certain antibody responses. Available preclinical data indicates that BG9588 does not cause a global blockage of the immune response to pathogens and that its effects are reversible upon clearance from the systemic circulation. In this Phase I/II open-label, multiple-dose, multicenter study, 30 subjects with active proliferative lupus nephritis will receive 20 mg/kg BG9588 by IV infusion once every 14 days for three doses, and then once every 28 days for four doses for a total of 7 doses. The primary objective is to determine if BG9588 can decrease proteinuria by greater than or equal to 50 percent from baseline without worsening renal function. The secondary objectives are to determine the safety and pharmacokinetics of BG9588, as well as the effects of BG9588 on renal flares; cellular casts; C(3) levels and anti-dsDNA titers; requirement for prednisone; general lupus activity; and quality of life.

ELIGIBILITY:
Must give written informed consent prior to any testing under this protocol.

Must be 18 years or older, inclusive, at the time of informed consent.

Must have a renal biopsy showing active WHO Class III, IV, or mixed membranous and proliferative SLE GN, within the 5 years prior to the first dose of study drug.

Must have proteinuria of greater than or equal to 1.0 g/day at both the Day-27 and day-13 evaluations.

Must fulfill any one the following four criteria, at each of the two screening visits (i.e., Day-27 and Day-13):

Anti-dsDNA antibody greater than 2x the upper limit of normal (ULN).

C3 complement less than 80 mg/dL.

Hematuria greater than 5 rbc/hpf.

Urinary granular or red blood cell casts.

Must not have any medical disorder, which in the opinion of the investigator, should exclude the subject from this study.

Must not have prior arterial or venous thrombosis, or history of recurrent abortion (3 or more), in the presence of anti-cardiolipin antibodies.

Must not have a chest x-ray with evidence of active infection or neoplasm within the 6 months prior to the first dose of study drug.

Must not have rapidly progressive glomerulonephritis, defined as a doubling of serum creatinine, within the 3 months prior to the first dose of study drug.

Must not have fibrinoid necrosis and/or cellular crescents affecting more than 25 percent of glomeruli in any renal biopsy performed within the 3 months prior to the first dose of study drug.

Must not have clinically significant findings for any of the following within the 4 weeks prior to the first dose of study drug: active psychiatric disease, serum creatinine greater than 2.0 mg/dL, prothrombin time (PT) greater than 1.3x control (in the absence of coumadin therapy; abnormal PT values due to anti-coagulation therapy are allowed if within the therapeutic range), AST or ALT levels greater than 3x normal, other major organ dysfunction, or serious local or systemic infection (e.g., pneumonia, septicemia).

Must not be positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HVC Ab), or HIV antibody at the Day-27 evaluation.

Must not have a mean CD4 count less than or equal to 300 microliters (mean of Day-27 and Day-13 results).

Must not have treatment with an antibody or other investigational drug within the 3 months prior to the first dose of the study drug.

Must not have any vaccination within the 4 weeks prior to the first dose of the study drug.

Must not have treatment with IV or oral cyclophosphamide within the 4 weeks prior to the first dose of the study drug.

Must not have treatment with any of the following medications within the 4 weeks prior to the first dose of study drug: IV methylprednisolone, cyclosporine or related compound, or oral prednisone (equivalent oral glucocorticoid) at a dose greater than 0.5 mg/kg/day.

Must not have initiation of treatment with ACE inhibitors within the 4 weeks prior to the first dose of study drug.

Must not have initiation of treatment with azathioprine, methotrexate or mycophenolate mofetil within the 4 weeks prior to the first dose of study drug.

Must not have treatment with any new oral or new IV antibiotic within the 2 weeks prior to the first dose of study drug. Subjects on prophylactic antibiotics are permitted to continue these during the study.

Female subjects, unless post-menopausal or surgically sterile, must use an adequate method of contraception.

Women must not be currently breast-feeding.

Must not have a positive pregnancy test in any evaluation prior to the first dose of study drug.

Must not be currently enrolled in any other study in which the subject is receiving any type of drug or non-drug therapy.

Must not have been previously dosed with BG9588.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1999-06; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, Domenech I, Aydintug AO, Jedryka-Goral A, de Ramon E, et al. Systemic lupus erythematosus: clinical and immunologic patterns of disease expression in a cohort of 1,000 patients. The European Working Party on Systemic Lupus Erythematosus. Medicine (Baltimore). 1993 Mar;72(2):113-24. PMID 8479324